CLINICAL TRIAL: NCT06712992
Title: Effect of Trans-Spinal Direct Current Stimulation in the Management of Non-Specific Chronic Low Back Pain: A Randomized Controlled Trial
Brief Title: Electromyographic Response to TsDcs in CNSLBP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: German International University (Other)
Responsible Party: Principal Investigator, Ahmed Medhat Mahfouz Elgamal, Principal invistigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T/REC/2024.10021
Record Dates: First submitted 2024-11-26; First posted 2024-12-03 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trans-spinal direct current stimulation group (Experimental): Patients in this group will receive Conventional Exercises in addition to tsDCS. We will apply a current density of 0.035 mA/cm2 and will deliver a total charge density of 42.8 mC/cm2, below the threshold values reported for tissue damage. For tsDcs, At the onset of tsDCS, the current will be increased for 30 s, and at the offset, it will be decreased for 30 s in a ramp-like manner. Participants will receive three sessions of treatment per week for four weeks, with a total of twelve sessions.
  Interventions: Device: Trans-spinal Direct Current Stimulation; Other: Conventional Exercises
- Sham Trans-spinal direct current stimulation group (Sham Comparator): Patients in this group will receive Conventional Exercises in addition to SHAM tsDCS. For a sham tsDCS, the current will be ramped up for 30 seconds turned on for 5 s and then turned off in a ramp shaped fashion, thus inducing skin sensations indistinguishable from anodal tsDCS. This method was shown to achieve a good level of blinding among sessions. Participants will receive three sessions of treatment per week for four weeks, with a total of twelve sessions.
  Interventions: Other: Conventional Exercises; Drug: SHAM Trans-spinal Direct current stimulation

INTERVENTIONS:
Device: Trans-spinal Direct Current Stimulation — Physiomed- IONOSON-Expert, Germany will be used to deliver SHAM direct current, The Physiomed- IONOSON-Expert, Germany is Two-channel electrotherapy including 21 currents, including direct current. The tsDCS electrodes will be rectangular pieces of saline-soaked synthetic sponge (7 × 8 cm, 56 cm2), to minimize chemical reactions at the electrode-skin interface. The anode will be placed over the spinous process of the eighth thoracic vertebra (T8) and the cathode will be placed on the second lumbar vertebra (L2) according to a modeling study which demonstrated that this configuration had a relevant impact on the distribution of the induced electric field (EF) in the lumbosacral spinal cord for the efficacy of tsDCS.
  Arms: Trans-spinal direct current stimulation group
Other: Conventional Exercises — 1. Isometric exercises of spine
     * Hollowing in abdominals.
     * Isometric for back extensors.
  2. Bridging exercises.
  3. Graded active flexion exercises of spine
  4. Graded active extension exercises of spine
Drug: SHAM Trans-spinal Direct current stimulation — For a sham tsDCS, the current will be ramped up for 30 seconds turned on for 5 s and then turned off in a ramp shaped fashion, thus inducing skin sensations indistinguishable from anodal tsDCS. This method was shown to achieve a good level of blinding among sessions.
  These parameters for sham stimulation were chosen based on previous reports that the perceived sensations on the skin, such as tingling, fade usually out in the first 30 s of TsDcs .
  Arms: Sham Trans-spinal direct current stimulation group

SUMMARY:
The purpose of this randomized, double-blinded, sham-controlled study is to investigate the efficacy of trans-spinal direct current stimulation on pain level, quality of life, and electromyographic nociceptive flexion reflex in patients with non-specific chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both sexes.
* Age 18-60 years old.
* Chronic non-specific low back pain according to the most recent guidelines for the diagnosis and management of NSLPB come from the American College of Physicians and was published in 2017. According to these guidelines, the diagnosis of chronic NSLBP should be made based on the following criteria:
* Chronic low back pain, defined as pain lasting for more than 12 weeks.
* No specific identifiable cause of pain(e.g. infection, malignancy, fracture, inflammatory disorder).
* No radicular symptoms(e.g. pain radiating down the leg).
* No significant neurological deficits or findings on physical examination(e.g. loss of reflexes or muscle strength).

Exclusion Criteria:

* Previous fractures and/or surgery in the vertebral spine.
* Neuropathic pain extending along the lower limb due to nerve root compression.
* History of spine trauma or fracture.
* Implanted pacemakers.
* Pregnancy.
* Malignancy.
* Systemic musculoskeletal diseases.
* Epilepsy.
* History of psychiatric disorders.
* Obesity

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-10 (Estimated)

PRIMARY OUTCOMES:
Changes in NPRS from baseline to four weeks | Baseline and 4 weeks
  An 11-point Numerical Pain Rating Scale (NPRS; 0= no pain, 10= maximum pain) will be used to assess the patients' pre and post treatment levels of back pain. The NPRS can be administered verbally (therefore also by telephone) or graphically for self-completion. Scores range from 0-10 points, with higher scores indicating greater pain intensity

SECONDARY OUTCOMES:
Changes in Nociceptive Flexion Reflex (NFR) Threshold and area from baseline to 4 weeks | Baseline and 4 weeks
  The NFR threshold will be assessed as an objective measure of spinal nociceptive processing in adults with chronic non-specific low back pain (CNSLBP). The NFR threshold will be defined as the lowest stimulus intensity that elicits an NFR response.The NFR threshold and NFR area will be assessed before and after 4 weeks of trans-spinal direct current stimulation (tsDCS) plus exercise or sham stimulation plus exercise.
Changes in PROMIS Global Health - 10 Survey from baseline to 4 weeks | Baseline and 4 weeks
  The Patient-Reported Outcomes Measurement Information System (PROMIS) is a comprehensive instrument designed to assess health-related quality of life across various domains. PROMIS GH-10, specifically, is tailored to measure global physical and mental health. It encompasses a range of items that evaluate general health perceptions, physical function, pain, fatigue, emotional distress, and social health. PROMIS GH-10 has been demonstrated to be reliable and valid for use in the general population and various specific conditions, such as low back pain.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Sixth of October, Giza Governorate
  - Outpatient clinical of faculty of physical therapy, Ahram Canadian University, Sixth of October, Giza Governorate

IPD SHARING:
Plan to Share IPD: No